CLINICAL TRIAL: NCT01715480
Title: Physiological Effect of Sulforaphane Obtained From Broccoli Sprouts Homogenates (BSH) on the HbF and Anti-oxidative Capacity of Human Sickle Red Blood Cells (SS RBC)
Brief Title: Effect of Broccoli Sprouts Homogenate on SS RBC
Acronym: BSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00033630
Record Dates: First submitted 2012-03-06; First posted 2012-10-29 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-02

CONDITIONS: Sickle Red Blood Cell; Fetal Hemoglobin; Oxidative Stress
Keywords: broccoli sprout; sickle cell; NRF2
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Broccoli sprout homogenate ingestion (Experimental): Subjects will ingest broccoli sprout homogenate in the form of a shake.
  Interventions: Dietary Supplement: Broccosprouts® (Brassica Protection Products LLC) homogenate

INTERVENTIONS:
Dietary Supplement: Broccosprouts® (Brassica Protection Products LLC) homogenate — In the in-vitro part of the study, sulphoraphane will be added into the culture media used to grow and differentiate the erythroid cells from blood samples obtained from three Hb AA volunteers and three Hb SS subjects. The subjects will have a single clinic visit for the blood donation.
  In the second part of the study, enrolled subjects will be asked to consume homogenates of broccoli sprouts by mouth daily for three weeks. They will have a maximum of five clinic visits for medical assessments and lab draws during this time. They will then have a final clinic visit after a washout period of six weeks.
  Other Names: Broccoli sprout

SUMMARY:
The overall purpose of this study is to obtain a better understanding of the biological response of red blood cells to sulforaphane contained in fresh broccoli sprouts that have been put through a blending process. This study will use commercially available fresh broccoli sprouts certified by Brassica Protection Products LLC (BroccoSprouts®). This product can also be purchased at some local grocery stores in the produce section. It is believed that NRF2, a transcription factor encoded by the NFE2L2 gene, plays a role in the regulation of defense against oxidative stress. The detrimental accelerated breakdown of sickle cell disease (SCD) red blood cells (SS RBC) is partially due to reduced anti-oxidative capacity. Previous analysis of SS RBC microRNAs revealed that a reduced level of NRF2, the master regulator of anti-oxidative stress capacity, contributes to reduced resistance to oxidative stress and increased hemolysis; NRF2 also induces fetal hemoglobin (HbF), which is known to prevent SS RBC sickling.

First, erythroid progenitors from normal and SCD subjects will be tested ex-vivo to find out how sulforaphane, a natural NRF2 activator, affects the oxidative stress capacity, HbF expression, and microRNA expression of red cells.

Second, a pilot clinical trial will be conducted to determine the safety and physiological effects of 3 weeks of daily consumption of broccoli sprout homogenate in a cohort of Hb SS/SB0 thalassemia adult SCD patients. During this study, subjects RBCs will be assayed for changes in anti-oxidative stress capacity and microRNA composition in mature SCD red blood cells.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hemoglobin (Hb) SS or Hb Sβ0 thalassemia by electrophoresis
* Age ≥18 years
* Hematocrit (Hct) ≥ 20% and Hb > 6.0 g/dL
* Capacity to understand and sign informed consent and can adhere to the daily regimen of BSH

Exclusion Criteria:

* RBC transfusion or change in hydroxyurea dose during the 3 months prior to study entry
* Ongoing pregnancy
* Diabetes
* Renal insufficiency (BUN >21 mg/dL and/or Creatinine >1.4 mg/dL)
* History of allergy to sulfonamides

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2012-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
In vitro response of HbAA and HbSS erythroid cells to NRF2 activation by sulforaphane. | 3 months
  Erythroid progenitor cells from 3 volunteers with Hb AA and 3 subjects with Hb SS disease will be exposed to sulforaphane and then their expression levels of genes regulated by Nrf2 will be measured.
Safety, physiological effects and cellular effects of daily consumption of broccoli sprout homogenate in a cohort of Hb SS/SB0 thalassemia adult SCD patients | 1-2 years
  Adult subjects with Hb SS/SB0 thalassemia will be recruited to participate in this part of the study. Subjects will be asked to consume broccoli sprout that have been blended into a milkshake-like substance daily for three consecutive weeks. Safety measures will include recording of vital signs and adverse signs and symptoms. Assessment of physiological effects will include measurement of blood chemistries, counts, LDH, and hemoglobin F level. Measurements of cellular effects will include changes in microRNA gene profiling, gene expression profiling, and quantitation of anti-oxidant capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Jen-Tsan A Chi, MD, PhD, Principal Investigator — Duke University; Marilyn J Telen, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Background] Sangokoya C, Telen MJ, Chi JT. microRNA miR-144 modulates oxidative stress tolerance and associates with anemia severity in sickle cell disease. Blood. 2010 Nov 18;116(20):4338-48. doi: 10.1182/blood-2009-04-214817. Epub 2010 Aug 13. PMID 20709907
- [Derived] Doss JF, Jonassaint JC, Garrett ME, Ashley-Koch AE, Telen MJ, Chi JT. Phase 1 Study of a Sulforaphane-Containing Broccoli Sprout Homogenate for Sickle Cell Disease. PLoS One. 2016 Apr 12;11(4):e0152895. doi: 10.1371/journal.pone.0152895. eCollection 2016. PMID 27071063